CLINICAL TRIAL: NCT04442399
Title: Pilot of Family-based Self-management for HIV-infected Adolescents in Two Clinics in Ndola
Brief Title: Family Connection: Pilot of Family-based Self-management for HIV-infected Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00006271
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2020-06

CONDITIONS: HIV; Adolescent Behavior; Caregivers; Africa
Keywords: HIV; Adolescents; Youth; Caregivers; Africa; Intervention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention was based on the WHO-endorsed manual entitled Positive Connections: Leading Information and Support Groups for Adolescents Living with HIV. For Family Connections, a caregiver companion guide was developed. In brief, adolescent/caregiver pairs attended 10 intervention sessions held every other Saturday at their HIV clinic over a six-month period.
  Interventions: Behavioral: Family Connections
- Comparison (No Intervention): The comparison arm consisted of standard of care for adolescents as offered at the HIV clinics.

INTERVENTIONS:
Behavioral: Family Connections — Ten intervention sessions were covered, ranging form understanding HIV and to handling stigma and discrimination.
  Arms: Intervention

SUMMARY:
The study design has two phases. The first phase is the refinement of intervention manual for an adolescent living with HIV (ALHIV)and their caregiver intervention, followed by a second phase feasibility pilot study. The study goals are to refine and pilot a feasible intervention that fosters resiliency and draws upon the strengths of adolescents and their families. Specific aims include to: (1) Refine activities and an intervention manual for a family-focused group intervention for adolescents and their caregivers to improve HIV self-management among adolescents living with HIV; (2) conduct a pilot study to assess the acceptability and feasibility of the group intervention among 50 adolescent/caregiver pairs that are randomly assigned to the intervention or the comparison arms, and (sub aim 2a) examine preliminary trends in outcome measures, including Anti-Retroviral Therapy (ART) adherence, safer sex behaviors and stigma, comparing the intervention and comparison study arms.

DETAILED DESCRIPTION:
The need for effective interventions to support adolescent HIV self-management is particularly pressing in Sub-Saharan Africa (SSA) where the majority of the 2.1 million ALHIV reside. Highlighting the vulnerability of ALHIV is their increasing HIV-related mortality, up 50% in 2012 compared to 2005, while the global number of HIV-related deaths among all ages decreased by 30%. In response to the disparate burden of HIV mortality among ALHIV, combined with the compelling evidence from HIV prevention and chronic illness literature and research on the influential role of families, the study team propose to refine and pilot test an ALHIV/caregiver group intervention. This intervention will draw upon principles of Positive Youth Development (PYD) and Social Cognitive theory (SCT) to emphasize skills building, self-efficacy, youth participation, and strengthening adult relationships. The intervention will build upon an existing ALHIV support group guide and utilize trained facilitators to hold group sessions with ALHIV and their caregivers to: 1) improve understanding of HIV among ALHIV and caregivers; 2) help ALHIV develop strategies for healthy living including adherence to ART; 3) build the capacity of ALHIV to make informed decisions about their sexual and reproductive health; 4) build the capacity of caregivers to support ALHIV; and 5) help ALHIV develop life skills to communicate their HIV diagnosis effectively, and to plan for their future. The study design has two phases. The first phase is the refinement of the ALHIV/caregiver intervention manual followed by a second phase feasibility pilot study. The Study goals are to refine and pilot a feasible intervention that fosters resiliency and draws upon the strengths of adolescents and their families. Specific aims include to: (1) Refine activities and an intervention manual for a family-focused group intervention for adolescents and their caregivers to improve HIV self-management among adolescents living with HIV; (2) conduct a pilot study to assess the acceptability and feasibility of the group intervention among 50 adolescent/caregiver pairs that are randomly assigned to the intervention or the comparison arms, and (sub aim 2a) examine preliminary trends in outcome measures, including ART adherence, safer sex behaviors and stigma, comparing the intervention and comparison study arms.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents: 15 and 19 years old, aware of their HIV status, and had been on ART for at least six months
* Caregivers:nominated by the adolescents and were at least 20 years old

Exclusion Criteria:

- Caregiver: Being a biological parent is not an eligibility criterion

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of adolescent/caregiver pairs who attend Family Connections (feasibility) | Attendance over the course of the 6 month intervention collected using attendance log.
  Feasibility was assessed based on attendance at the intervention sessions.We considered the intervention feasible if at least two-thirds of the pairs attended 80% or more of the intervention sessions.
Proportion of participants who would recommend the Family Connections program (acceptability) | At the six-month endline data collection
  The proportion of participants who reported during the endline survey that they would recommend the intervention to others.

SECONDARY OUTCOMES:
Youth Participants' mean ART adherence over six months using daily medication electronic monitoring system (MEMS) caps data | Collected monthly over the course of the six month intervention
  Medication electronic monitoring system (MEMS) caps data recorded the date and time the pill bottle was opened.
Proportion of participants with viral failure (1,000 copies or more per mL) | ~ 6 months (from baseline to endline)
  Defined as having 1,000 or more RNA copies per mL
Youth Participants' adolescent internalized stigma measures (yes/no) | ~ 6 months (from baseline to endline]
  Three agree/disagree statements from the Internalized AIDS Stigma Scale (IA-RSS) as adapted previously in Zambia - low chronbach's alpha resulted in the three measures being analyzed as separate indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Denison, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Ndola, Zambia

IPD SHARING:
Plan to Share IPD: No
We did not get assent/consent from participants to make their data available to a third party, therefore we are not able to make the data publicly available, rather our consent forms specified the following "the study research team will have access to your data. This team includes the study investigators, research assistants and data analysts".